CLINICAL TRIAL: NCT03167905
Title: Comparison of the Role of Epidural Analgesia Versus Non-epidural Analgesia in Postnatal Depression and Persistent Pain Development: a Randomized Controlled Trial
Brief Title: CODEPAD (Collaborative Outcomes of DEpression and Pain Associated With Delivery)
Acronym: CODEPAD
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/2090
Record Dates: First submitted 2017-05-02; First posted 2017-05-30 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Depression, Postpartum; Analgesia, Obstetrical; Anesthesia, Obstetrical
Keywords: Anesthesia, Obstetrical; Epidural anesthesia; Postnatal depression; Persistent pain
MeSH Terms: conditions — Depression, Postpartum; Agnosia | interventions — Entonox; Nitrous Oxide; Meperidine; Remifentanil; Fentanyl; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Cross over or switch to the other group of analgesia is allowed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural group (Experimental): Patients are assigned to receive epidural delivery system (fentanyl and ropivacaine) for labour as pain relief option.
  Interventions: Device: Epidural delivery system; Drug: Fentanyl; Drug: Ropivacaine
- Non-epidural group (Active Comparator): Patients are assigned to receive entonox (laughing gas), meperidine (pethidine) or remifentanil (Ultiva) for labour as pain relief option.
  Interventions: Drug: Entonox; Drug: Meperidine; Drug: Ultiva

INTERVENTIONS:
Device: Epidural delivery system — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Arms: Epidural group
Drug: Entonox — Entonox will be given upon request in non-epidural group.
  Other Names: Laughing gas
  Arms: Non-epidural group
Drug: Meperidine — Intramuscular pethidine (75mg/1.5ml) will be given upon request in non-epidural group.
  Other Names: Pethidine
  Arms: Non-epidural group
Drug: Ultiva — Intravenous patient controlled remifentanil (20-40mcg/ml) is only given when the patient rejects or cannot receive pethidine and entonox in non-epidural group..
  Other Names: Remifentanil
  Arms: Non-epidural group
Drug: Fentanyl — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Arms: Epidural group
Drug: Ropivacaine — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Arms: Epidural group

SUMMARY:
Postnatal depression affects about 10-15% of women after childbirth. Approximately 3-5% of women experience a moderate-to-severe depression that requires medical attention. This study aims to investigate the implication of pain relief choice in reducing the postnatal depression of women who deliver their babies.

DETAILED DESCRIPTION:
If the patients have not decided on which pain relief method to be used, and would like to take part in this study, they will be assigned to either epidural or non-epidural pain relief for labour based on the study randomization result. Blood samples will be drawn to study the presence of known functional polymorphisms in candidate genes associated with depression, pain, stress and anxiety. Patients will be followed up with study questionnaires related to pain and postnatal depression screening during the study. For some of the patients, a discrete choice experiment (DCE) on pain relief choice will be conducted, and their preferences on epidural analgesia will be asked.

During any time of the labour period, the patient is allowed to switch the pain relief option upon request.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (American Society of Anesthesiologists physical status 1 and 2) parturients at term (36 weeks gestation or more) (nulliparous and multiparous);
* With a singleton fetus.

Exclusion Criteria:

* Multiple pregnancies;
* Non-cephalic fetal presentation;
* Obstetric complications (e.g. pre-eclampsia, uncontrolled hypertension, uncontrolled diabetes);
* Elective and urgent caesarean section (not from delivery suite).

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 881 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of major postnatal depression in both groups | 6-10 weeks after delivery
  Edinburgh Postnatal Depression Scale (EPDS) score>=13
The incidence of (clinically significant, probable) postnatal depression in both groups | 6-10 weeks after delivery
  Edinburgh Postnatal Depression Scale (EPDS) score>=10

SECONDARY OUTCOMES:
The incidence of acquiring post-delivery persistent pain in both groups | 6-10 weeks after delivery
  Pain score>3 in the perineal, surgical scar or abdomen region that lasts for at least 6 weeks post-delivery
Pain vulnerability in both groups (1) | Upon recruitment until 6-10 weeks after delivery
  Assessment via Pain Catastrophizing Scale (PCS) questionnaire before and after delivery
Pain vulnerability in both groups (2) | Upon recruitment until 6-10 weeks after delivery
  Assessment via Central Sensitisation Inventory (CSI) questionnaire before and after delivery
Pain vulnerability in both groups (3) | Upon recruitment till end of first stage of labor (1 day)
  Assessment via Angle Labor Pain Questionnaire (A-LPQ) during first stage of labor when the participants experience labor pain
Psychological vulnerability in both groups (1) | Upon recruitment until 5 days after delivery
  Assessment via Fear-Avoidance Components Scale (FACS) questionnaire before delivery
Psychological vulnerability in both groups (2) | Upon recruitment until 5 days after delivery
  Assessment via State Trait Anxiety Inventory (STAI) questionnaire before delivery
Psychological vulnerability in both groups (3) | Upon recruitment until 5 days after delivery
  Assessment via Perceived Stress Scale (PSS) questionnaire before delivery
Pain severity in both groups | During labour till one day after delivery
  Pain score>3 during labour
Preferences for labor analgesia | Prior to labor and delivery
  Recruited patients will be administered a survey on Discrete Choice Experiment (DCE) and other questions on their preferences for labor analgesia. For DCE, nine tasks will be included in which parturients will choose one of four hypothetical forms of labor analgesia: 1) epidural analgesia, 2) pethidine, 3) Entonox (nitrous oxide-oxygen mixture), and 4) no labor analgesia, which varies with regards to six attributes: 1) pain intensity following treatment, 2) duration of second stage of labor, 3) risk of instrumental delivery, 4) risk of back pain, 5) risk of permanent nerve injury, and 6) out-of-pocket cost.
Preferences for epidural analgesia | Prior to labor and delivery
  Recruited patients will be administered a survey on their preferences and opinions on epidural analgesia, including their concerns on possible risk of epidural analgesia e.g. instrumental delivery, prolonged duration of second stage of labor, back pain etc.
Chinese version of Angle Labor Pain Questionnaire (A-LPQ) | Upon recruitment till end of first stage of labor (1 day)
  Assessment via Angle Labor Pain Questionnaire (A-LPQ) during first stage of labor when the participants experience labor pain. The tool comprises 22 items divided into five subscales on the childbirth pain experience: the enormity of the pain, the fear and anxiety, uterine contraction pain, birthing pain, and the back pain/ long haul. Each item is scaled from 0 to 10, implying a range from non to worst possible or extremely (where applicable), and therefore has a total score ranged from 0 to 220. The higher the score, the greater the labor pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan HS, Tan CW, Sultana R, Chen HY, Chua T, Rahman N, Gandhi M, Sia ATH, Sng BL. The association between epidural labour analgesia and postpartum depression: a randomised controlled trial. Anaesthesia. 2024 Apr;79(4):357-367. doi: 10.1111/anae.16178. Epub 2023 Nov 21. PMID 37990597
- [Derived] Chan JCY, Sultana R, Mathur D, Tan CW, Sng BL. The association of pain and psychological vulnerabilities with postpartum pain catastrophizing: a secondary analysis of a randomized controlled trial. Can J Anaesth. 2025 Apr;72(4):603-614. doi: 10.1007/s12630-025-02920-8. Epub 2025 Mar 20. PMID 40113655
- [Derived] Ayuby NA, Ang MQ, Sultana R, Tan CW, Sng BL. Investigating the association between labor pain and cessation of breastfeeding. Sci Rep. 2024 Dec 28;14(1):31361. doi: 10.1038/s41598-024-82850-5. PMID 39732915
- [Derived] Tan CW, Tan NY, Sultana R, Tan HS, Sng BL. Investigating the association factors of acute postpartum pain: a cohort study. BMC Anesthesiol. 2023 Jul 25;23(1):252. doi: 10.1186/s12871-023-02214-w. PMID 37491196
- See also: Published data on the primary outcome on epidural labour analgesia and postnatal depression — https://pubmed.ncbi.nlm.nih.gov/37990597/